CLINICAL TRIAL: NCT05527938
Title: The Effectiveness of Web-based Interventions on Nonalcoholic Fatty Liver Disease (NAFLD) in Obese Children: A Study Protocol for a Randomized Controlled Trial
Brief Title: Web-based Interventions on Nonalcoholic Fatty Liver Disease (NAFLD) in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaoxing Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Xu Renjie, Pharmacist, Shaoxing Maternity and Child Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ShaoxingMaternityChildHC
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: NAFLD; Web; Childhood Obesity
Keywords: NAFLD; obese children; web; education; protocol
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: web-based intervention
Who Masked: Participant
Masking Description: Study personnel involved in the data assessment of the study are blinded to the patients' treatment assignment. The clinical doctors that deliver the study treatment are not blinded and are therefore uninvolved in the patients' data assessments related to this study. Data analysts are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- web-based intervention (Experimental): 1. Establishing management teams.
  2. Establishment of a nursing intervention team.
  3. Daily uploading of health intervention records
  4. Regularly delivering related health knowledge.
  5. Home visiting
  6. Psychological guidance.
  Interventions: Other: web-based intervention
- the control group (No Intervention): 1. Routine care.At each visit to the hospital, in this time, the child and his parents are given health education on diet and exercise booklets, and the parents supervise the child's daily life.
  The team members will review the child's condition every month for feedback.

INTERVENTIONS:
Other: web-based intervention — 1. Establishing management teams.
  2. Establishment of a nursing intervention team.
  3. Daily uploading of health intervention records
  4. Regularly delivering related health knowledge.
  5. Home visiting
  6. Psychological guidance. The health teachers in the team should closely understand the psychological trends of the patients during the telephone follow-up and home visits and verbally communicate more with the children to stimulate them to develop good living habits and increase their confidence in healing.
  Arms: web-based intervention

SUMMARY:
The web-based continuity of care intervention model to provide comprehensive nursing interventions for obese children with NAFLD, always tracking their performance status, enabling them to grasp the knowledge of healthy weight loss, develop good lifestyle habits, and reduce their weight, thus reducing the incidence of NAFLD in children.

DETAILED DESCRIPTION:
The web-based continuity of care intervention model to provide comprehensive nursing interventions for obese children with NAFLD, always tracking their performance status, enabling them to grasp the knowledge of healthy weight loss, develop good lifestyle habits, and reduce their weight, thus reducing the incidence of NAFLD in children.The primary outcome are serum biomarkers such as alanine aminotransferase (ALT) and gamma-glutamyl transferase (GGT) . Second outcomes are: aspartate aminotransferase, and liver imaging (liver ultrasound and magnetic resonance imaging), BMI, waist-to-hip ratio and quality of life. In addition, socio-demographic characteristics such as age, gender and ethnicity will be recorded. All outcomes were measured at baseline, week 4, week 16, week 24, week 36, and week 48 to determine the trajectory of change in outcome variables over intervention process.

ELIGIBILITY:
Inclusion Criteria:

* The clinical diagnosis of Nonalcoholic Fatty Liver Disease

Exclusion Criteria:

* Patients do not agree to participate
* participate in other health intervention programs now

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The change of alanine aminotransferase（ALT）and gamma-glutamyl transferase（GGT） | Change from Baseline ALT and GGT at 48 weeks
  The primary outcome are serum biomarkers such as alanine aminotransferase (ALT) and gamma-glutamyl transferase (GGT) .

SECONDARY OUTCOMES:
The change of aspartate aminotransferase | Change from Baseline aspartate aminotransferase at 48 weeks
  Second outcome is aspartate aminotransferase
The change of liver imaging | Change from Baseline liver imaging at 48 weeks
  Third outcome is liver imaging
The change of BMI | Change from Baseline BMI at 48 weeks
  Fourth outcome is BMI
The change of waist-to-hip ratio | Change from Baseline waist-to-hip ratio at 48 weeks
  Fifth outcome is waist-to-hip ratio
The change of quality of life | Change from Baseline quality of life at 48 weeks
  Sixth outcome is quality of life

OTHER OUTCOMES:
socio-demographic characteristics such as age, gender and ethnicity | baseline
  In addition, socio-demographic characteristics such as age, gender and ethnicity will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Caixia Tian, MSc, Principal Investigator — Shaoxing Maternity and Child Health Care Hospital
Locations (1):
- Caixia Tian, Shaoxing, Zhejiang, China

REFERENCES:
- [Derived] Tian C, Xu J, Wang G, Yu L, Tang X. The effectiveness of web-based interventions on non-alcoholic fatty liver disease (NAFLD) in obese children: A study protocol for a randomized controlled trial. Front Public Health. 2022 Oct 20;10:930901. doi: 10.3389/fpubh.2022.930901. eCollection 2022. PMID 36339187